CLINICAL TRIAL: NCT05077722
Title: PISTACHIO (Preemption Of Disruptive Behavior In Children) Real-Time Monitoring Of Sleep And Behavior Of Children 3-7-Year-Old Receiving Parent Child Interaction Therapy Augmented With Artificial Intelligence Randomized Controlled Trial
Brief Title: Monitoring of Sleep and Behavior of Children 3-7 Years Old Receiving Parent-Child Interaction Therapy With the Help of Artificial Intelligence
Acronym: PISTACHIo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-007403
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Disruptive Behavior; Attention-deficit Hyperactivity; Oppositional Defiant Disorder
Keywords: Emotional Behavioral Dyscontrol
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Parent Child Interaction Therapy (Experimental): Subjects enrolled in Parent Child Interaction Therapy (PCIT) will wear a Garmin smartwatch that will provided targeted messages during tantrums picked up by the Garmin devices that will instruct them on how to deescalate their child.
  Interventions: Device: Garmin
- Sham Biometric - Parent Child Interaction Therapy (Sham Comparator): Subjects enrolled in Parent Child Interaction Therapy will wear Garmin smartwatch and will receive only random messages throughout the day with various relaxation strategies such as reminders to practice deep breathing with their child.
  Interventions: Device: Garmin

INTERVENTIONS:
Device: Garmin — A smartwatch device that measures subjects level of activity, heartrate, respirations and quality of your sleep at night. Artificial intelligence will be applied to analyze all the data over the course of 12 weeks to monitor and attempt to predict the onset of tantrums or disruptive behavior. Subjects are required to wear the watch at least 70% of the day and night each day for 70% of days during 12 weeks of treatment.

SUMMARY:
The purpose of this study is to develop an innovative wearable tracking protocol that will use Artificial Intelligence (AI) technology to monitor sleep and behavior of 3-7 year old children.

ELIGIBILITY:
Inclusion Criteria - Children:

* Ages 3-7.
* Outpatients or Inpatients.
* Any gender, race or ethnicity.
* Able to provide developmentally appropriate informed assent, and legal guardians able to provide informed consent .
* EBP Severity rated above the clinically significant range (≥120; T-score ≥ 60) (Eyberg Child Behavior Inventory- ECBI; Eyberg & Pincus, 1999).
* Need for more intensive behavioral treatments such as ER visit for behavioral dyscontrol or hospitalization will not be exclusionary or exit criteria.
* Families approached for participation will be asked to commit to complete the treatment.
* At least one primary caregiver and the identified child will have to be able to speak and understand English.

Exclusion Criteria - Children:

* Formal diagnosis of Severe Intellectual disability, Autistic Spectrum Disorder Level 3, or a psychotic disorder for the child.
* Parents not consenting to the study.
* Parents or child is not able to adhere to the study protocol.
* A Child who is reasonable expected to be unable to tolerate wearing the Garmin device for at least 70% of the time during the day and night 70% of the days during the treatment (12 weeks). This is based on the principal investigator's discretion.
* Unable to speak and understand English.
* Refusal or withdrawal of consent, inability, or unwillingness to adhere to study procedures.
* Children in foster care.

Inclusion Criteria - Adults:

* Agree to wear Garmin watch.
* Ages 18-99.
* Any gender, race, ethnicity.
* Able to provide informed consent.

Exclusion Criteria - Adults:

* Unable to speak and understand English.
* Refusal or withdrawal of consent, inability, or unwillingness to adhere to study procedures.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Garmin use | 12 weeks
  Number of days participants wear the Garmin smartwatch

SECONDARY OUTCOMES:
Eyberg Child Behavior Inventory | 12 weeks
  The Eyberg Child Behavior Inventory questionnaire is measured on two subscales for a series of phrases that describe a children's behavior. The first subscale is for indicating the frequency of the behavior using a scale of 1= never to 7 = Always; the second subscale indicates yes = 1 or no = 0 for whether the behavior is currently a problem for them. Reponses are total with a higher score indicating greater severity of child's behavior.
Pediatric Sleep Questionnaire | 12 weeks
  Pediatric Sleep Questionnaire to assess child's sleep with a series of 22 questions on a yes/no problem scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Croarkin, DO, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Romanowicz M, Saliba MT, Wilton AR, Garzon Hincapie JF, Croarkin KS, Saliba CT, LeMahieu A, Drapeau N, Schlichting B, Skime M, Bobo WV, Vande Voort JL, Shekunov J, Croarkin PE, Athreya AP. Feasibility of Digital Augmentation of Parent-Child Interaction Therapy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2548869. doi: 10.1001/jamanetworkopen.2025.48869. PMID 41396603
- [Derived] Saliba M, Drapeau N, Skime M, Hu X, Accardi CJ, Athreya AP, Kolacz J, Shekunov J, Jones DP, Croarkin PE, Romanowicz M. PISTACHIo (PreemptIon of diSrupTive behAvior in CHIldren): real-time monitoring of sleep and behavior of children 3-7 years old receiving parent-child interaction therapy augment with artificial intelligence - the study protocol, pilot study. Pilot Feasibility Stud. 2023 Feb 9;9(1):23. doi: 10.1186/s40814-023-01254-w. PMID 36759915
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials